CLINICAL TRIAL: NCT07315945
Title: Implementation of an Allergic Rhinitis Severity Questionnaire in ENT Consultations
Acronym: QSRA-ORL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9692
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; SCST score; SNOT 22 score
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Allergic rhinitis is a very common condition (affecting 1 in 5 people in Europe) and a costly one for society (direct and indirect costs). Symptoms vary depending on the time of year, and treatments are primarily symptomatic, with follow-up in ENT consultations. Scientific societies (EAACI, FDA, EMA) recommend using a universal tool (severity score) (the CSMS score, SCST in French) to monitor severity and follow-up, and to obtain consistent data that can be extrapolated to other scientific data (meta-analyses).

Therefore, investigators in the ENT department use this SCST score (as well as others such as the SNOT 22 score) to assess the severity of allergic rhinitis in our patients and its progression.

Tbe investigators wish to confirm the acceptability of this tool for patients, and the statistical value of its properties.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Follow-up at the ENT department of Hautepierre University Hospital for allergic rhinitis

Exclusion Criteria:

* Asymptomatic individuals not requiring follow-up consultations.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) having follow-up at the ENT department of Hautepierre University Hospital for allergic rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Self-Assessment Clinical Symptom Score (SCST) | Up to 6 months
  1. Rating Scale
     Each symptom is rated by the patient according to its intensity:
     * 0: absent
     * 1: mild
     * 2: moderate
     * 3: severe
  2. Calculating the Score
     * Add the scores for each symptom.
     * The total SCST score reflects the overall severity of the symptoms:
       * Low score → mild symptoms
       * High score → severe symptoms
  3. Interpretation
     * Before treatment: establish a baseline.
     * After treatment: compare the scores to assess effectiveness.
     * A decrease in the score indicates clinical improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France